CLINICAL TRIAL: NCT01546675
Title: Interface Kinematics of Transhumeral Prosthetic Sockets Using XROMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Lifespan (Other); Brown University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A9227-P
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Amputation of Arm
Keywords: Amputation; Prosthesis Design; Biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional 1, Skeletal Stabilization 2 (Active Comparator): Subjects using the Traditional Socket and socket hypothesized to increase skeletal stabilization in a case cross-over design. The intervention is the socket designed to increase skeletal stabilization.
  Interventions: Other: Skeletal Stabilization
- Skeletal Stabilization 1, Traditional 2 (Experimental): Subjects using the socket hypothesized to increase skeletal stabilization and Traditional Socket and in a case cross-over design. The intervention is the socket designed to increase skeletal stabilization.
  Interventions: Other: Skeletal Stabilization

INTERVENTIONS:
Other: Skeletal Stabilization — Upper Limb Prosthetic Socket hypothesized to increase skeletal stabilization
  Other Names: Skeletal Stabilization Socket

SUMMARY:
The purpose of this pilot study was to conduct a head-to-head comparison of two designs for transhumeral level upper limb prosthetic sockets: a traditional socket design and a socket design hypothesized to provide greater skeletal stabilization. The investigators comparisons included assessments of patient comfort and satisfaction with fit, as well as dynamic kinematic assessment using X-Ray Reconstruction of Moving Morphology (XROMM) a novel high-speed, high-resolution, bi-plane video radiography system.

DETAILED DESCRIPTION:
In the past decade, advances in upper limb socket design and technology have been proposed to increase comfort and decrease perceived weight of the prosthesis. There have been no scientific studies to date that have evaluated the benefits of these designs, and thus no evidence to support use of one type of prosthetic socket design over another. Thus, the overall purpose of this pilot study was to conduct a head-to-head comparison of two designs for transhumeral level upper limb prosthetic sockets: a traditional socket design and a socket design hypothesized to provide greater skeletal stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female transhumeral amputees, 18 years or older of any ethnicity, who are current prosthetic users.

Exclusion Criteria:

* Subjects with frozen shoulder of the residual side, and/or severely limited active range of motion of the shoulder joint of the residual limb
* Inability to tolerate wearing of a prosthetic socket
* Mental impairment that renders a subject unable to comply with the study
* Skin conditions such as burns or poor skin coverage as well as those with severe contractures that prevent prior prosthetic wear
* Any electrically controlled medical device including pacemaker, implanted defibrillator or drug pumps
* Neuropathy, uncontrolled diabetes, receiving dialysis
* Any other significant comorbidity which would interfere with the study
* Severe circulatory problems including peripheral vascular disease and pitting edema will be excluded
* Cognitive deficits or mental health problems that would limit ability to participate fully in the study protocol
* Women who are pregnant or who plan to become pregnant in the near future

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Resnik, PhD MS, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

REFERENCES:
- [Derived] Resnik L, Patel T, Cooney SG, Crisco JJ, Fantini C. Comparison of transhumeral socket designs utilizing patient assessment and in vivo skeletal and socket motion tracking: a case study. Disabil Rehabil Assist Technol. 2016;11(5):423-32. doi: 10.3109/17483107.2014.981876. Epub 2014 Nov 26. PMID 25425411

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Traditional 1, Skeletal Stabilization 2: Subjects using the Traditional Socket in the first 2 weeks and then the socket hypothesized to increase Skeletal Stabilization in the second two weeks in a case cross-over design.
- Experimental: Skeletal Stabilization 1, Traditional 2: Subjects using the Skeletal Stabilization Socket in the first 2 weeks and then the Traditional Socket in the second two weeks in a case cross-over design.
Period: Overall Study
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross-over design. Each subject participated under each condition. Total of 2 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2 | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 20 [20 to 20] | 29 [29 to 29] | 24.5 [20 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Degrees of Shoulder Abduction Within the Prosthetic Socket
Description: Shoulder abduction was performed to the subject's maximum elevation. Skeletal and socket kinematics were calculated using the markerless auto-registration algorithm and X-Ray Reconstruction of Moving Morphology (XROMM)
Time Frame: After 4 weeks of home use (2 weeks for each socket style)
Population: One male and one female with traumatic amputation at the transhumeral level.
Measure: Number; unit: degrees
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
degrees
  Skeletal Stabilization Socket | 27 | 23.7
  Traditional Socket | 42.5 | 20.3

2. Secondary Outcome: Trinity Amputations and Prosthetics Experience Satisfaction Scale (TAPES)
Description: This 10 item scale includes items related to satisfaction with aspects of the prosthesis. It includes questions about extent of satisfaction regarding functional characteristics of the artificial limb: reliability, comfort, fit, and overall satisfaction, contentment with cosmetic characteristics of the device. Each item is rated on a 5 point scale from very dissatisfied to very satisfied. Scores are summed and the average of the 10 items are calculated. Higher scores indicate greater satisfaction. Scores range from 1-5.
Time Frame: After 4 weeks of home use (2 weeks for each socket style)
Measure: Number; unit: units on a scale
Groups:
- Active Comparator: Traditional 1, Skeletal Stabilization 2: .Subjects using the Traditional Socket in the first 2 weeks and then the socket hypothesized to increase Skeletal Stabilization in the second two weeks in a case cross-over design.
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
units on a scale
  Skeletal Stabilization Socket | 2.7 | 3.2
  Traditional Socket | 3.4 | 5

3. Secondary Outcome: Prosthetic Evaluation Questionnaire (PEQ) - Utility Subscale
Description: The 8-item utility subscale includes items related to prosthetic socket utility including: comfort, fit, ease of donning and doffing and feel on the residual limb. All items were scored using a 1 to 7 Likert scale average with lower scores indicated worse ratings and higher scores indicated better ratings. The scores for each item were added and the total score was the average of scores for all items, thus scores could range from 1 to 7.
Time Frame: after 2 weeks of home use of each socket type
Measure: Number; unit: units on a scale
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
units on a scale
  Skeletal Stabilization Socket | 3.4 | 4.3
  Traditional Socket | 5.4 | 6.6

4. Primary Outcome: Degrees of Shoulder Internal Rotation Within the Prosthetic Socket
Description: Isometric internal rotation was performed with the prosthetic elbow flexed to 90 degrees and shoulder in neutral position. Skeletal and socket kinematics were calculated using the markerless auto-registration algorithm and X-Ray Reconstruction of Moving Morphology (XROMM)
Time Frame: After 4 weeks of home use (2 weeks for each socket style)
Measure: Number; unit: degrees
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
degrees
  Skeletal Stabilization | 17.1 | 5.9
  Traditional Socket | 14.1 | 21.6

5. Primary Outcome: Degrees of Shoulder Displacement Within the Prosthetic Socket
Description: A shoulder shrug task was achieved by pulling up on a strap attached to the load cell, which was mounted on the vertical face of the concrete pedestal. Skeletal and socket kinematics were calculated using the markerless auto-registration algorithm and X-Ray Reconstruction of Moving Morphology (XROMM)
Time Frame: After 4 weeks of home use (2 weeks for each socket style)
Measure: Number; unit: degrees
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
degrees
  Skeletal Stabilization Socket | 4.4 | 5.3
  Traditional Socket | 3.1 | 37.0

6. Secondary Outcome: Prosthetic Evaluation Questionnaire (PEQ) - Residual Limb Health Subscale
Description: The 6-item residual limb health scale includes items about the bothersome of sweating, smell, swelling, ingrown hairs, rashes and blisters. All items were scored using a 1 to 7 Likert scale average with lower scores indicated worse ratings and higher scores indicated better ratings. The scores for each item were added and the total score was the average of scores for all items, thus scores could range from 1 to 7.
Time Frame: After 4 weeks of home use (2 weeks for each socket style)
Measure: Number; unit: units on a scale
Arm/Group | Active Comparator: Traditional 1, Skeletal Stabilization 2 | Experimental: Skeletal Stabilization 1, Traditional 2
Number analyzed (Participants) | 1 | 1
units on a scale
  Skeletal Stabilization Socket | 4.7 | 5.5
  Traditional Socket | 6.2 | 4.7

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected during each participants study duration.
Groups:
- Cases: Subjects using the Traditional Socket and socket hypothesized to increase skeletal stabilization in a case cross-over design.
Arm/Group | Cases
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
These results cannot be generalized outside of this small sample and may have been different if the intervention socket had been optimized. Additional research is needed to expand our understanding of the impact of prosthetic socket designs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes